CLINICAL TRIAL: NCT06679504
Title: Quality of Life After Laparoscopic Totally Extraperitoneal Inguinal Hernia Repair With Fibrin Glue Versus Tack Mesh Fixation
Brief Title: Laparoscopic Totally Extraperitoneal Inguinal Hernia Repair With Fibrin Glue Versus Tack Mesh Fixation
Status: Completed | Type: Observational
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Waleed Ghareeb, Consultant and lecturer of Surgery, Suez Canal University
Other Study IDs: #4846/2022
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibrin glue group: Laparoscopic Totally Extraperitoneal Inguinal Hernia Repair With Fibrin Glue
  Interventions: Procedure: Fibrin glue fixation
- Tack fixation group: Laparoscopic Totally Extraperitoneal Inguinal Hernia Repair With Fibrin Glue Versus Tack Mesh Fixation
  Interventions: Procedure: Tack fixation

INTERVENTIONS:
Procedure: Fibrin glue fixation — Laparoscopic Totally Extraperitoneal Inguinal Hernia Repair With Fibrin Glue fixation
  Groups: Fibrin glue group
Procedure: Tack fixation — Laparoscopic Totally Extraperitoneal Inguinal Hernia Repair With Tack Mesh Fixation
  Groups: Tack fixation group

SUMMARY:
The quality of life after hernia surgery like chronic pain and discomfort has frequently been reported with a frequency varying from 0 to 53%. As many as 10% of the patients report increased pain following surgery. Therefore, the current study aimed to assess the quality-of-life for patients with post-inguinal hernia repair by mesh fixation versus fibrin glue.

DETAILED DESCRIPTION:
A wide variety of mesh fixation techniques are available for laparoscopic hernia repair. These can be broadly divided into mechanical and nonmechanical methods. Mechanical methods include sutures and tissue penetrating fixation devices like tackers. Nonmechanical techniques include self-gripping meshes and tissue adhesives (glues).

Mechanical methods are hypothesized to cause more postoperative pain and increased risk of seroma formation, hematoma formation, and osteitis pubis due to tissue trauma and also have increased risk of chronic pain due to nerve entrapment. On the other hand, nonmechanical methods do not have these disadvantages.

Furthermore, the quality of life after hernia surgery like chronic pain and discomfort has frequently been reported with a frequency varying from 0 to 53%. As many as 10% of the patients report increased pain following surgery. Such a chronic pain is often developed due to the use of open inguinal technique along with heavy weight mesh with mechanical fixation techniques, presence of severe pain before surgery and young age. To the best of our knowledge, there are lacking evidence assessing the impact of mesh fixation using fibrin glue upon the quality of life of patients. Therefore, the current study aimed to assess the quality-of-life for patients who had post inguinal hernia repair by mesh fixation versus fibrin glue.

ELIGIBILITY:
Inclusion Criteria:

1. Age group of 18-60 years.
2. All types of inguinal hernias.
3. Didn't undergo pervious hernia repair surgery.

Exclusion Criteria:

1. Patients who are unfit for general anesthesia or with American Society of Anesthesiologists (ASA) grade 3 and above.
2. Presence of other groin or abdominal hernias.
3. Patients with complicated hernias such as irreducibility, obstruction, and incarceration.
4. Patients with obesity or morbid obesity BMI >= 35.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients complain of uncomplicated inguinal hernia who are scheduled for laparoscopic TEP hernioplasty
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of life assessment | 7 days, 15 days, 1 month, 2 months, and 3 months.
  The postoperative quality of life has been compared between both groups using SF-36 scoring questionnaire. The SF-36 is a 36 item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). The higher scores mean better quality of life..

SECONDARY OUTCOMES:
Postoperative pain assessment | 7 days, 15 days, 1 month, 2 months, and 3 months.
  VAS; visual analogue scale. for pain assessment. the score ranges from 1-10... higher score denotes more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Tolba, PhD, MD, Study Director — Suez canal University Hospital
Locations (1):
- Suez Canal University, Ismailia, Egypt